CLINICAL TRIAL: NCT04972825
Title: Autism Intervention Network for Behavioral Health- Mind the Gap
Brief Title: AIR-B4: Mind the Gap
Acronym: MTG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Collaborators: University of Rochester (Other); University of Kansas (Other); University of Pennsylvania (Other); Drexel University (Other); University of California, Davis (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Connie Kasari, Ph.D., Professor of Human Development and Psychology, Health Resources and Services Administration (HRSA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-001403
Record Dates: First submitted 2021-07-01; First posted 2021-07-22 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Autism Spectrum Disorder; Neurodevelopmental Disorders
Keywords: new diagnosis; autism services; Mind the Gap; navigating program
MeSH Terms: conditions — Autism Spectrum Disorder; Neurodevelopmental Disorders | interventions — mtg protein, Drosophila

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UNITED (Experimental): UNITED is premised on the idea that successful implementation in organizations like schools and early intervention systems requires a team-based approach, in which the team is thoughtfully assembled, develops a plan for implementation, assigns roles and responsibilities, and carefully tracks and supports implementation and sustainment in all its stages within a few meetings and ongoing coaching from the research staff.
  Interventions: Behavioral: Mind the Gap
- Implementation as Usual (IAU) (Active Comparator): The organizations will implement Mind the Gap as usual. The research team will be available to provide support on the Mind the Gap intervention as needed.
  Interventions: Behavioral: Mind the Gap

INTERVENTIONS:
Behavioral: Mind the Gap — This intervention will help parents with children newly diagnosed with autism or other neurodevelopmental disorders learn how to navigate the system of acquiring services for their child. These parents will be assisted by a coach, an employee at the child's agency, that will help them through this process.

SUMMARY:
The AIRB research team will compare the use and effectiveness of each intervention (Mind the Gap, Remaking Recess and Self Determination Learning Model of Instruction) with and without the addition of an implementation strategy, UNITED. In all groups, the research team will train community practitioners using remote delivery of professional development modules specific to the intervention, and active coaching for up to 12 sessions as dictated by the intervention procedures during a time span of 6 months.

The research team will pair UNITED with three interventions that cover the ages of early childhood, childhood, and adolescence. These include Mind the Gap (MTG), a family navigation intervention for children newly diagnosed under age 8, Remaking Recess (RR), a school-based social/peer engagement intervention for children ages 5-12, and Self-Determination Learning Model of Instruction (SDMLI), a self-advocacy intervention for adolescents (13-22 years; 22 is the upper age limit of high school for individuals with disabilities).

For MTG, peer navigators (staff working in an organization that already works with parents) and parents (with children with ASD) will meet via phone or video conference for up to 12 sessions within a 6 month span (an hour each time). They will go over sessions that were created by the research group that help parents understand the system of acquiring services. The total time commitment for peer navigators is about 18 hours and for parents with children with ASD is about 8.5 hours.

Identified families connected to the community organization will be matched with one peer navigator who will then guide and support the caregiver through completion of the MTG modules with active coaching of the family. Family needs and preferences will guide topic selection. Active coaching will occur via zoom, or over the phone, based on family preference and some recorded sessions will be shared with the research group for analyses. Mind the Gap will be available in English, Spanish, and Korean.

DETAILED DESCRIPTION:
Mind the Gap will include 20 agency staff, 48 Peer Navigators working at participating community organizations with peer navigator capacity (e.g. parent support centers; FQHC; community clinics; faith-based agencies) serving children with ASD and other NDD; and 240 families of children age 2-8 (with potential expansion based on community feedback) with ASD or NDD.

Training will be provided by experts in each intervention at each CRE. MTG targets peer navigators (parents of children with disabilities) who will complete the 12- hour remote training on MTG modules and associated topics (e.g., boundaries, family and child safety, data collection). The research team will conduct the initial 12 hours of training and active coaching/check ins during the 12 sessions the peer navigator has with the family in a 6-month span. Agency staff (supervisors or managers of agencies) will be also be given the training to help facilitate the training of the peer navigators at their respective sites and participate in UNITED if randomized to receive it. Identified families connected to the community organization will be matched with one peer navigator who will then guide and support the caregiver through completion of the MTG modules with active coaching of the family. Family needs and preferences will guide topic selection. Active coaching will occur via zoom, or over the phone, based on family preference.Consents can be signed online via Qualtrics, DocuSign (UC Davis) or RedCap for the parents, peer navigators, and agency staff. The parents participating in Mind the Gap will fill out a Demographic, Family Empowerment Scale, Permission to Contact, and WHO QOL Scale at entry. They will also fill out the following surveys at exit (6 months): Family Empowerment Scale and Caregiver Satisfaction Survey. Mind the Gap will be available in English, Spanish, and Korean. Peer navigators will fill out the following surveys at entry after signing consent: demographic, implementation climate scale, and social network surveys. They will also fill out surveys at 12 months and 18 months, which consist of social network surveys, implementation climate scale and an exit survey (only at 12 months).

All participants in Mind the Gap will be randomized to receive UNITED, exploratory implementation strategy, or implementation as usual (IAU). UNITED is premised on the idea that successful implementation in organizations like schools and early intervention systems requires a team-based approach, in which the team is thoughtfully assembled, develops a plan for implementation, assigns roles and responsibilities, and carefully tracks and supports implementation and sustainment in all its stages. To address these requirements, we combine two well- tested strategies. The first is social network analysis (SNA) through which we will systematically identify members of the team who will implement each intervention. The second is TeamSTEPPS (Team Strategies and Tools to Enhance Performance and Patient Safety), an evidence-based set of teamwork tools that optimizes target population outcomes by improving communication and teamwork skills. The research staff will approach the site leaders (2 at maximum) at agencies and explain MTG. After the site leaders agree to participate in the study, they will complete an agency agreement to participate and then fill out the Social Network Assessment (SNA) to provide names, roles, and emails of staff at the agency that have significant roles in the agency that relate to the Mind the Gap intervention. The research staff will then email these agency staff the SNA as well. After receiving the completed SNA assessments, we will randomize each organization to UNITED vs Implementation as Usual (IAU). We will use the data from these assessments to assess both arms of the study. Additionally, for those randomized to UNITED, Dr. Elizabeth McGhee Hassrick at Drexel University and her team, will provide the research sites the top 2-5 agency staff identified by the SNA as key for intervention implementation support. This team will be invited to participate in the UNITED implementation team. If they agree, they will complete an Agency Rep Consent before beginning any UNITED training. For both UNITED and IAU sites, peer navigators will be recruited from the agency based on leader recommendations. They will complete the Peer Navigator Consent prior to beginning Mind the Gap training.

ELIGIBILITY:
Inclusion Criteria:

* families of children age 2 to 8 with ASD or NDD. no receipt of ASD specific services outside of school (family may still qualify if child is connected with a regional center/EI, but not yet receiving services), defined as (a) services obtained through insurance based on having an ASD diagnosis; or (b) receiving services through 0-3 that can only be accessed with an ASD dx (e.g., intensive in home EIBI); (3) family income is under 250% of the federal guidelines for poverty rate; (4) English, Korean or Spanish speaking.
* agency staff (coordinators, directors, managers, supervisors) working on community organizations with peer navigator capacity e.g. parent support centers; FQHC; community clinics; faith-based agencies) serving children with ASD and other NDD (neurodevelopment disorders).
* peer navigators which include people working at participating community organizations with peer navigator capacity (e.g. parent support centers; FQHC; community clinics; faith-based agencies) serving children with ASD and other NDD (neurodevelopment disorders)

Exclusion Criteria:

* families with children under the age of 2 or over 8 years of age, does not have ASD or NDD; parents are not fluent in English, Spanish, or Korean; child already receiving services accessed with an ASD diagnosis; family income is over 250% federal guidelines for poverty rate
* Agency Staff: people not working in an organization that has a peer navigator capacity; cannot commit to the requirements of the study.
* Peer Navigators: people not working in an organization that has a peer navigator capacity; cannot commit to the times and requirements of the study

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2021-07-29 (Actual); Primary Completion 2025-12-23 (Estimated); Study Completion 2026-01-05 (Estimated)

PRIMARY OUTCOMES:
Stages of Implementation Completion (SIC) | through study completion, an average of 18 months
  Tool developed by the Oregon Social Learning Center, is an 8 stage tool of implementation process and milestones, with stages spanning three implementation phases (pre-implementation, implementation, and sustainability. The research staff will enter dates once milestones are completed.

SECONDARY OUTCOMES:
School Implementation Climate Scale (SICS) | baseline (entry), 12 months, and 18 months
  This scale was adapted to be used by the research team to gather information from the schools/agencies in the study about the use of evidence-based practices in their organizations. It is rated from 0 to 4, with 0 being "not at all" and 4 being "very great extent." The higher the rating, the better the outcome.
Change in Coaching Session Data Form from month to month | monthly from baseline and up to 6 months after baseline
  This form was created within the research group. It is used monthly after entry to document the services the participants would like to get and the ones they are currently receiving.
Family Empowerment Scale (Koren, DeChillo & Friesen, 1992) | baseline and 6 months
  It is a 34-item rating scale that measures empowerment in families with children who have emotional, behavioral, or developmental disorders. The FES has three subscales, Family, Service System and, Social Politics. Parents rated each item on a 5-point Likert-type rating scale. It is rated from 1 to 5, with "1" being never and "5" being very often. The higher the rating, the better the outcome.
WHOQOL scale | baseline
  Adapted from WHOQOL -BREF Questionnaire, to gather information about the quality of life and health from the families in the study. It is rated from 0 to 5, with "0" being not at all and "5" being completely. The higher the rating, the better the outcome.
Social Network Survey | baseline, 12 months, and 18 months
  Survey created by the research team to gather information about the key people in each organization that can better support the Mind the Gap intervention.
Caregiver Satisfaction Survey | 6 months after baseline
  This survey was created by the research team. At 6 months post entry, caregivers will rate their satisfaction with the intervention on a survey that utilizes a 5-point Likert-type rating scale.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UC Davis MIND Institute, Davis, California
  - University of Kansas, Lawrence, Kansas
  - University of Rochester, Rochester, New York
  - UPENN, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Locke J, Hassrick EM, Stahmer AC, Iadarola S, Boyd B, Mandell DS, Shih W, Hund L, Kasari C; AIR-B Network. Using Novel Implementation Tools for Evidence-based Intervention Delivery (UNITED) across public service systems for three evidence-based autism interventions in under-resourced communities: study protocol. BMC Psychiatry. 2022 Jul 16;22(1):478. doi: 10.1186/s12888-022-04105-9. PMID 35842614